CLINICAL TRIAL: NCT04188509
Title: An Open-Label Extension Study of Voxelotor Administered Orally to Participants With Sickle Cell Disease Who Have Participated in Voxelotor Clinical Trials
Brief Title: Open-Label Extension of Voxelotor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-038; 2019-003144-76 (EudraCT Number); C5341023 (Other: Alias Study Number)
Expanded Access: NCT04724421 (No longer available)
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Intervention Model Description: Open-Label Extension study available to eligible participants from GBT-sponsored voxelotor clinical studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor (Experimental): All participants will receive voxelotor once daily (QD), administered orally as tablets, dispersible tablets, or a stick pack formulation (powder blend formulation packaged as stick packs). Participants aged ≥ 12 years and/or ≥ 40 kgs will receive a voxelotor dose of 1500 mg QD. Participants aged < 12 years and < 40 kgs will receive weight based dosing of voxelotor. The participant's weight at study entry will be used to determine the starting voxelotor dose in this study. Participants may receive study drug as long they continue to receive clinical benefit that outweighs risk as determined by the investigator and/or until the participant has access to voxelotor from an alternative source.
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — All participants will receive voxelotor once daily (QD), administered orally as tablets, dispersible tablets, or a powder for oral suspension formulation (powder formulation packaged as stick packs).
  Other Names: GBT440

SUMMARY:
Open-label extension study of voxelotor for participants with Sickle Cell Disease who have participated in voxelotor clinical trials.

DETAILED DESCRIPTION:
Open-label extension (OLE) study of voxelotor for participants with Sickle Cell Disease who have participated in voxelotor clinical trials. Up to approximately 600 participants with sickle cell disease (SCD), will be enrolled at approximately 70 clinical sites globally. All participants will receive voxelotor once daily, administered orally as tablets, dispersible tablets, or powder for oral suspension formulation. The objective of this OLE is to assess the safety of, and SCD-related complications of, long-term treatment with voxelotor, in participants who have completed treatment in a Global Blood Therapeutics (GBT)-sponsored voxelotor clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant with SCD, who participated and received study drug in a GBT-sponsored voxelotor clinical study.

Note: Participants who discontinued study drug due to an AE, but who remained on study, may be eligible for treatment in this study provided the AE does not pose a risk for treatment with voxelotor.

Note: Participants who discontinued Study GBT440-032 as the result of an abnormal transcranial Doppler (TCD) flow velocity assessment (≥ 200 cm/sec) are eligible for treatment in this study.

- Participant has provided written consent/assent (for pediatric participants, both the consent of the participant's legal representative or legal guardian and the participant's assent [where applicable] must be obtained).

Exclusion Criteria:

* Female participant who is breastfeeding or pregnant
* Participant withdrew consent from a GBT-sponsored voxelotor clinical study
* Known hypersensitivity to voxelotor or any other components of the study drug
* Use of St. John's wort, sensitive cytochrome P450 (CYP) 3A4 substrates with a narrow therapeutic index, or moderate or strong CYP3A4 inducers within 30 days of Day 1

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (6):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta Scottish Rite, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Missouri
  - ECU Physicians, Brody Outpatient Clinic, Greenville, North Carolina
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Egypt (4):
  - Zagazig University Hospital, Zagazig, Alsharkia
  - Alexandria University Hospital - Clinical Research Center, Alexandria
  - Cairo University Hospital, Abu El Rish Hospital, Cairo
  - Ain Shams University Hospital - Clinical Research Center (MASRI-CRC), Cairo
- Lebanon (2):
  - American University of Beirut - Medical Center, Beirut
  - Nini Hospital, Tripoli
- Nigeria (5):
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - College of Medicine, University of Ibadan, Ibadan, Oyo State
  - Barau Dikko Teaching Hospital/Kaduna State University, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos
- United Kingdom (3):
  - University College Hospital NHS Foundation Trust, London, Greater London
  - Barts Health NHS Trust , The Royal London Hospital, London
  - Guy'S and St Thomas' Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-038

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 162 participants who had previously completed the following studies: GBT440-032 (NCT04218084) who received placebo, and GBT440-007 (NCT02850406), GBT440-032 (NCT04218084) or GBT440-042 (NCT05561140) who received voxelotor were enrolled in the study GBT440-038 (NCT04188509). All participants enrolled in this study received voxelotor.
Groups:
- Voxelotor: Participants aged >= 12 years received voxelotor 1500 milligrams (mg) once daily (QD) tablets. Participants aged < 12 years received a voxelotor dose based on their body weight to provide exposure corresponding to the adult dose of 1500 mg QD as powder for oral suspension or dispersible tablet or modified dispersible tablet. Participants received study drug as long they continued to receive clinical benefit that outweighed risk as determined by the investigator and/or until the participant had access to voxelotor from an alternative source.
Period: Overall Study
Arm/Group | Voxelotor
Started | 162
Completed | 25
Not Completed | 137
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal of Consent | 1
Not completed — Discretion of Investigator | 1
Not completed — Noncompliance | 3
Not completed — Sponsor Decision | 127
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Voxelotor: Participants aged >= 12 years received voxelotor 1500 mg QD tablets. Participants aged < 12 years received a voxelotor dose based on their body weight to provide exposure corresponding to the adult dose of 1500 mg QD as powder for oral suspension or dispersible tablet or modified dispersible tablet. Participants received study drug as long they continued to receive clinical benefit that outweighed risk as determined by the investigator and/or until the participant had access to voxelotor from an alternative source.
Arm/Group | Voxelotor
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.2 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 161
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 94
  Race: Arab | 2
  Race: Black or African American | 40
  Race: Middle Eastern or North African | 9
  Race: White | 10
  Race: Multi-Racial | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered to be drug related. A treatment emergent AE was defined as an AE with an onset date on or after the date of informed consent until 28 days after discontinuation of drug. AEs included both serious AEs (SAEs) and all non-SAEs. An SAE was an AE or suspected adverse reaction that, at any dose, in the view of the either the investigator or sponsor, resulted in any of the following outcomes: death, was life-threatening, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From date of informed consent until 28 days after last dose of study drug (maximum up to 4.31 years)
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Voxelotor
Number analyzed (Participants) | 162
Participants | 105

2. Primary Outcome: Number of Participants With SAEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered to be drug related. An SAE was an AE or suspected adverse reaction that, at any dose, in the view of the either the investigator or sponsor, resulted in any of the following outcomes: death, was life-threatening, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From date of informed consent until 28 days after last dose of study drug (maximum up to 4.31 years)
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Voxelotor
Number analyzed (Participants) | 162
Participants | 53

3. Primary Outcome: Number of Participants With Sickle Cell Disease (SCD) Related TEAEs and SAEs
Description: SCD-related AEs were common complications associated with the study participant's SCD and were not considered to be related to voxelotor unless judged by the investigator to have worsened in severity and/or frequency or changed in nature during the study. SCD-related complications included the following: sickle cell anemia with crisis, acute chest syndrome (ACS), pneumonia, priapism, and osteonecrosis. A treatment emergent AE was defined as an AE with an onset date on or after the date of informed consent until 28 days after discontinuation of drug. An SAE was an AE or suspected adverse reaction that, at any dose, in the view of either the investigator or sponsor, resulted in any of the following outcomes: death, was life-threatening, resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From date of informed consent until 28 days after last dose of study drug (maximum up to 4.31 years)
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Voxelotor
Number analyzed (Participants) | 162
Participants
  SCD related treatment emergent AE | 60
  SCD related SAEs | 43

ADVERSE EVENTS:
Time Frame: From date of informed consent until 28 days after last dose of study drug (maximum up to 4.31 years)
Description: Same events may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. The safety population included all participants who received at least one dose of study drug.
Arm/Group | Voxelotor
All-Cause Mortality (participants affected / at risk) | 1/162
Serious Adverse Events (participants affected / at risk) | 53/162
Other Adverse Events (participants affected / at risk) | 93/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voxelotor (N=162)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 35 (75)
Anaemia (Blood and lymphatic system disorders) | 16 (41)
Splenic sequestration crisis (Blood and lymphatic system disorders) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Haemolysis (Blood and lymphatic system disorders) | 1 (2)
Urethral valves (Congenital, familial and genetic disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 8 (9)
Non-cardiac chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Malaria (Infections and infestations) | 8 (8)
Sepsis (Infections and infestations) | 6 (9)
Pneumonia (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 3 (3)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1)
Acute haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (2)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 15 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voxelotor (N=162)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 27 (53)
Anaemia (Blood and lymphatic system disorders) | 9 (12)
Thrombocytosis (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Splenic sequestration crisis (Blood and lymphatic system disorders) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Cholesteatoma (Ear and labyrinth disorders) | 1 (1)
Vernal keratoconjunctivitis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (11)
Vomiting (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 20 (32)
Non-cardiac chest pain (General disorders) | 3 (7)
Decreased activity (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 2 (2)
Jaundice (Hepatobiliary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 13 (25)
Malaria (Infections and infestations) | 10 (11)
Gastroenteritis (Infections and infestations) | 5 (5)
Influenza (Infections and infestations) | 5 (6)
COVID-19 (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 4 (7)
Viral infection (Infections and infestations) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (6)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3)
Adenovirus infection (Infections and infestations) | 1 (1)
Body tinea (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Mumps (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin candida (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Platelet count increased (Investigations) | 5 (5)
Eosinophil count increased (Investigations) | 4 (4)
Red cell distribution width abnormal (Investigations) | 3 (3)
Blood calcium decreased (Investigations) | 2 (2)
Blood urea decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Mean cell volume decreased (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (9)
Cluster headache (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1)
Painful erection (Reproductive system and breast disorders) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Splenectomy (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04188509/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04188509/SAP_001.pdf